CLINICAL TRIAL: NCT04536714
Title: Stress and Depression: Interventional, Non-pharmaceutical Stress Management Program With the Cognitive Restructuring Method "Pythagorean Self-Awareness" for Patients Diagnosed With Major Depressive Disorder
Brief Title: Efficacy of Pythagorean Self-Awareness Intervention for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evgenia E. Psarraki (Other)
Responsible Party: Sponsor-Investigator, Evgenia E. Psarraki, MSc, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prot.1 26/8/2020
Record Dates: First submitted 2020-08-26; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder
Keywords: major depression; stress management program
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 34 participants. Received Pythagorean Self-Awareness program
  Interventions: Behavioral: Pythagorean Self-Awareness Intervention program
- Control group (No Intervention): 35 participants. Received usual care

INTERVENTIONS:
Behavioral: Pythagorean Self-Awareness Intervention program — Stress management program of Pythagorean Self-Awareness Intervention (PSAI), which included eight sessions and lasted for eight weeks. On the first week, a personal session took place for measurements and training in the relaxation technique of diaphragmatic breathing. In the second week, patients attended a group session, in which they were adviced to follow specific directions for a healthy lifestyle, such as organized physical activity, adherence to the Mediterranean diet, creating a daily routine. In the third week, participants were introduced to the cognitive restructuring technique of (PSAI).In the following four group sessions, patients were trained on PSAI and the second relaxation technique, progressive muscular relaxation. In the last week, the final measurements were made. All sessions lasted for 120 minutes, except for the final one, which lasted for 60 minutes.
  Arms: Intervention group

SUMMARY:
The present study explored the effects of the implementation of the Pythagorean Self Awarenes Intervention (PSAI) on patients diagnosed with major depressive disorder. The primary aim was to evaluate the effectiveness of PSAI compared to the usual care provided for adults with major depressive disorder with respect to the reduction of depressive symptoms. Secondary aims of this study included reduction of stress and anxiety, enhancement of healthy lifestyle and improvement of affect, sleep quality and cognitive functions of patients.

DETAILED DESCRIPTION:
Study design This randomized controlled trial was conducted at the Mental Health Center of Peristeri, department of the Psychiatric Hospital of Attica, Greece, from December 2018 to January 2020. The study protocol was approved by the School of Medicine, National and Kapodistrian University of Athens (Protocol n. 1718038002/30/07/2018) and the center's directorate and was consistent with the Declaration of Helsinki. All participants were enlisted in the study only after being fully informed by the researcher about the aims and procedures of the research and submitting written consent.

Procedures Patients eligible for the above mentioned criteria were randomized in two groups: the intervention group, receiving PSAI, and the control group, receiving the usual care provided by the center for patients with MDD, namely medical treatment and counselling. Randomization was conducted based on random numbers generated by an online random number generator (https://www.sealedenvelope.com/simple-randomiser/v1/lists). This study was non-blinded, as patients and researchers were aware of the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder diagnosis conducted by a psychiatrist of the center according to the DSM-V criteria
* residency in Attica
* ability to speak and write fluently in the Greek language

Exclusion Criteria:

* antecedent psychotic or manic episode
* current feeding or eating disorder, obsessive-compulsive disorder, self-harming behaviors or recent suicide attempt and current drug abuse or addiction
* current treatment with Cognitive-Behavioral Therapy
* denial to participate in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | 2 months
  self-report questionnaire

SECONDARY OUTCOMES:
Healthy Lifestyle and Personal Control Questionnaire | 2 months
  self-report questionnaire
Depression-Anxiety-Stress Scale-21 | 2 months
  self-report questionnaire
Positive and Negative Affect Schedule | 2 months
  self-report questionnaire
Pittsburg Sleep Quality Index | 2 months
  self-report questionnaire
Brief International Assessment of Cognition for Multiple Sclerosis | 2 months
  battery of three cognitive tests
Hair cortisol concentration | 2 months
  Hair specimens from the posterior vertex of the scalp, three proximal to scalp cms
Salivary cortisol concentration | 2 months
  saliva specimens,three measurements in 24 hours: two in the morning (on awakening and 40 minutes later) and one at night (at 8:00). CAR and diurnal slope of cortisol were also calculated

CONTACTS AND LOCATIONS:
Overall Officials: Evgenia E Psarraki, MSc, Principal Investigator — MSc "The Science of Stress and Health Promotion", School of Medicine, NKU Athens; Christina Darviri, Dr, Study Director — MSc "The Science of Stress and Health Promotion", School of Medicine, NKU Athens
Locations (1):
- Mental Health Center of Peristeri, department of the Psychiatric Hospital of Attica, Ploutonos 19, Peristeri, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heim C, Binder EB. Current research trends in early life stress and depression: review of human studies on sensitive periods, gene-environment interactions, and epigenetics. Exp Neurol. 2012 Jan;233(1):102-11. doi: 10.1016/j.expneurol.2011.10.032. Epub 2011 Nov 7. PMID 22101006
- [Background] Hammen C. Stress and depression. Annu Rev Clin Psychol. 2005;1:293-319. doi: 10.1146/annurev.clinpsy.1.102803.143938. PMID 17716090
- [Background] Dean J, Keshavan M. The neurobiology of depression: An integrated view. Asian J Psychiatr. 2017 Jun;27:101-111. doi: 10.1016/j.ajp.2017.01.025. Epub 2017 Jan 29. PMID 28558878
- [Background] Winnebeck E, Fissler M, Gartner M, Chadwick P, Barnhofer T. Brief training in mindfulness meditation reduces symptoms in patients with a chronic or recurrent lifetime history of depression: A randomized controlled study. Behav Res Ther. 2017 Dec;99:124-130. doi: 10.1016/j.brat.2017.10.005. Epub 2017 Oct 12. PMID 29078199
- [Background] Wetherell JL, Hershey T, Hickman S, Tate SR, Dixon D, Bower ES, Lenze EJ. Mindfulness-Based Stress Reduction for Older Adults With Stress Disorders and Neurocognitive Difficulties: A Randomized Controlled Trial. J Clin Psychiatry. 2017 Jul;78(7):e734-e743. doi: 10.4088/JCP.16m10947. PMID 28686822
- [Background] Meyer B, Berger T, Caspar F, Beevers CG, Andersson G, Weiss M. Effectiveness of a novel integrative online treatment for depression (Deprexis): randomized controlled trial. J Med Internet Res. 2009 May 11;11(2):e15. doi: 10.2196/jmir.1151. PMID 19632969
- [Background] Rentala S, Fong TC, Nattala P, Chan CL, Konduru R. Effectiveness of body-mind-spirit intervention on well-being, functional impairment and quality of life among depressive patients - a randomized controlled trial. J Adv Nurs. 2015 Sep;71(9):2153-63. doi: 10.1111/jan.12677. Epub 2015 May 12. PMID 25967378
- [Background] Darviri, C., Zavitsanou, C., Delikou, A., Giotaki, A., Artemiadis, A., Terentiou, A., & Chrousos, G. P. (2016). A novel non-pharmaceutical treatment for patients with mild cognitive impairment. Psychology, 7(5), 678-686.
- [Background] Tsoli S, Vasdekis S, Tigani X, Artemiadis A, Chrousos G, Darviri C. A novel cognitive behavioral treatment for patients with chronic insomnia: A pilot experimental study. Complement Ther Med. 2018 Apr;37:61-63. doi: 10.1016/j.ctim.2018.01.015. Epub 2018 Feb 1. PMID 29609939
- [Background] Charalampopoulou M, Bacopoulou F, Syrigos KN, Filopoulos E, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on breast cancer patients undergoing adjuvant therapy: A pilot randomized controlled trial. Breast. 2020 Feb;49:210-218. doi: 10.1016/j.breast.2019.12.012. Epub 2019 Dec 20. PMID 31901782
- [Background] Darviri C, Alexopoulos EC, Artemiadis AK, Tigani X, Kraniotou C, Darvyri P, Chrousos GP. The Healthy Lifestyle and Personal Control Questionnaire (HLPCQ): a novel tool for assessing self-empowerment through a constellation of daily activities. BMC Public Health. 2014 Sep 24;14:995. doi: 10.1186/1471-2458-14-995. PMID 25253039
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Beck depression inventory-II. San Antonio, 78(2), 490-498.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Langdon DW, Amato MP, Boringa J, Brochet B, Foley F, Fredrikson S, Hamalainen P, Hartung HP, Krupp L, Penner IK, Reder AT, Benedict RH. Recommendations for a Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS). Mult Scler. 2012 Jun;18(6):891-8. doi: 10.1177/1352458511431076. Epub 2011 Dec 21. PMID 22190573
- [Background] Wester VL, van Rossum EF. Clinical applications of cortisol measurements in hair. Eur J Endocrinol. 2015 Oct;173(4):M1-10. doi: 10.1530/EJE-15-0313. Epub 2015 Apr 29. PMID 25924811
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637
- [Derived] Psarraki EE, Bacopoulou F, Panagoulias E, Michou M, Pelekasis P, Artemiadis A, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on patients with major depressive disorder: A pilot randomized controlled trial. J Psychiatr Res. 2021 Jun;138:326-334. doi: 10.1016/j.jpsychires.2021.03.067. Epub 2021 Apr 13. PMID 33894540